CLINICAL TRIAL: NCT04957264
Title: Assessment of Extubation Readiness in Preterm Infants Using Chest Ultrasound
Brief Title: Ultrasound for Assessment of Extubation Readiness
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0211-E
Record Dates: First submitted 2021-05-20; First posted 2021-07-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-10

CONDITIONS: Mechanical Ventilation Complication; Premature Birth
Keywords: Extreme preterm; neonates; Mechanical ventilation; Extubation, chest; Ultrasound
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preterm infants are at high-risk for the negative implications of both prolonged mechanical ventilation and extubation failure. Pre-extubation assessments of lung parenchyma and diaphragmatic function of these infants can be useful adjunctive tool for prediction of extubation readiness.

The aim of this study is to assess the sensitivity and specificity of lung ultrasound and diaphragmatic function evaluation in prediction of extubation readiness in mechanically ventilated neonates born at < 28 weeks gestational age.

DETAILED DESCRIPTION:
Study Design and setting:This is a prospective descriptive pilot study that will be conducted on infants born at < 28 weeks gestation who meet eligibility criteria and are admitted to the Neonatal intensive care at Mount Sinai Hospital. Enrolment of eligible infants will start after obtaining approval from Mount Sinai Research Ethics Board and parent's consent.

Time of assessment: Parents of infants on invasive mechanical ventilation who are eligible for the study will be approached for consent. Once the decision made by attending physician to extubate the infant, Chest ultrasound (Lung ultrasound + diaphragmatic function assessment) will be done. Chest ultrasound will be done before next feeding to avoid any interference of a full stomach on diaphragmatic assessment.

Study procedure: Decisions about extubation will be as per the clinical judgment of the physician in-charge of the infant and will not in any way based on Chest ultrasound measurements. A lung ultrasound combined with diaphragmatic function assessment will be done by one of the investigators prior to extubation. The result of Chest ultrasound will be masked for the clinical team to avoid any influence of the Chest ultrasound result on the extubation decision. On the other hand, if the attending physician requests Chest ultrasound for the purpose of the ongoing clinical management or to help with making extubation decision then the result of the study will be disclosed to the physician and this infant will be excluded from the study.

A random sample of 20% of eligible infants will have lung ultrasound scoring and diaphragmatic function assessment done twice by 2 operators (with various levels of Chest ultrasound expertise). None of the operator will be aware of the result of Chest ultrasound done by the other operator for the same patient. Lung ultrasound severity score, diaphragmatic thickness fraction and diaphragmatic excursion will be calculated. Inter-rater agreement will be assessed using raw percentage of agreement (Pa), Cohen's and Kappa (κ), and G wet agreement coefficient (AC1). Intra-class correlation will be determined for variables with continuous measurements (mixed factorial design). High-resolution linear and curvi-linear ultrasound probes of 20-5 and 10-3 MegaHertZ will be used to assess lung ultrasound score and to measure diaphragmatic thickness and diaphragmatic excursion [amplitude] respectively using both B-mode and M-mode.

Lung ultrasound assessment technique: Chest ultrasound will be performed in a standardized manner. A longitudinal scan of the anterior and lateral chest walls will be performed. Three chest areas for each side (upper anterior, lower anterior, and lateral) will be assessed. Each area will have a score of 0 to 4 points with the total score ranges from 0 to 24 which inversely correlating with lung aeration.

Diaphragmatic assessment technique: Diaphragm assessment will be performed in the supine position. For measuring diaphragmatic excursion, the curvilinear probe will be placed on the lower intercostal spaces between the mid-clavicular and anterior axillary lines on the right side. Using the B mode, the proper exploration line of the diaphragm will be detected by directing the beam perpendicular to the posterior third of each hemi-diaphragm. By M mode, the cyclic caudal diaphragmatic displacement with respiration will be measured as the perpendicular distance between the most caudal point of the liver or spleen at the end of expiration and the end of inspiration. The average of three respiratory cycles will be taken.

The assessment of the diaphragmatic efficiency as a pressure generator will be evaluated using the diaphragmatic thickness fraction. Diaphragmatic thickness will be measured at the apposition zone which can be obtained by placing the linear transducer above the 10th rib in the mid-axillary or anterior axillary lines in the right intercostal spaces. By B-mode, three distinct layers will be seen, the diaphragm as a hypo-echoic area bordered by two clear echogenic lines of the pleural membrane (upper line) and the peritoneal membrane (lower line). Using M-mode tracing, inspiratory diaphragmatic thickness will be measured as the maximum perpendicular distance between pleural and peritoneal layers and by the same way expiratory diaphragmatic thickness will be recorded. diaphragmatic thickness Fraction will be calculated using the following formula: diaphragmatic thickness Fraction equal to [(inspiratory thickness _ expiratory thickness)/expiratory thickness] x100. The average of the calculated diaphragmatic thickness Fraction from three respiratory cycles will be estimated. All Chest Ultrasound assessments will be undertaken using a standard aseptic technique.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are born at < 28 weeks Gestational Age,
* Admitted to the neonatal intensive care at Mount Sinai Hospital
* Receiving invasive mechanical ventilation.

Exclusion Criteria:

* Infants who are born at >27 weeks Gestational Age,
* On non-invasive mechanical ventilation
* Infants having congenital or chromosomal abnormalities,
* Infants intubated for < 12 hours
* Infants who have neurological insult, pneumothorax, or under muscle relaxant.
* If parents declined the consent.

Min Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants born at < 28 weeks Gestational Age, are admitted to the neonatal intensive care at Mount Sinai Hospital, and receiving invasive mechanical ventilation for at least 12 hours will be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of chest ultrasound in Prediction of extubation readiness in neonates born at less than 28 weeks gestation. | 2 year
  Chest ultrasound will be performed prior to extubation and Lung aeration will be scored based on three chest areas for each side (upper anterior, lower anterior and lateral) and a score of 0-to-4 point will be given for each area. The minimum score = 0 point and the maximum score = 24 points. successful extubation was defined as remained extubated at day 3 post extubation

SECONDARY OUTCOMES:
Assess the Diaphragmatic Thickness Fraction and Diaphragmatic Excursion in preterm infants | 2 year
  * Assessment of Diaphragmatic Thickness in millimetres.
  * Assessment of Diaphragmatic Excursion in millimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Mohamed, MD, Study Chair — Mount Sinai Hospital- Toronto, ON, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada